CLINICAL TRIAL: NCT01093248
Title: Methadone Maintenance Treatment Outcome Study in Taiwan
Acronym: M0508
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 99A1-PHPP39; 99A1-PHPP39 (Other Grant/Funding Number: National Health Research Institutes)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Heroin Addiction
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heroin-addicted Patients: Heroin-addicted outpatient department (OPD) patients who seek help for methadone maintenance treatment

SUMMARY:
Opioid abuse is a complex problem, which not only impacts on the affected individuals' physical and psychological health, but also threatens public security and the productivity of the society. Further, through needle sharing and sexual contacts, injecting drug users (IDUs) have become laden with HIV and HIV related health problems, representing a serious public health threat all over the world. In Taiwan, since the identification of the first HIV-infected IDU in 1987, the incident cases have continued to increase, reaching a height of 2,461 in 2005. In order to contain the epidemics of HIV among IDUs, and to prevent its spread to the population in general, the Center for Disease Control (CDC) collaborated with the Department of Justice to initiate and implement a number of harm reduction programs in 2005. The fact that opioid addiction is officially treated as a health rather than a legal issue itself represents a remarkable milestone in Taiwan. Among these harm reduction programs, including needle and syringe exchange for IDUs as well as substitution treatment approaches for opioid dependence, methadone maintenance treatment (MMT) perhaps represents the most most important and most crucial component. Remarkably, in a relatively short time span, more than 60 MMT programs were established, which enrolled more than 15,000 heroin addicts. This notwithstanding, the overall and differential effectiveness of these MMT service delivery systems, as well as the characteristics of these programs and the patients that might contribute toward treatment response or failure remain largely unknown. Such knowledge base is crucial for establishing standardized and feasible outcome evaluation processes for opioid addicts receiving MMT programs, as well as for the further improvement of the efficacy and effectiveness of these programs, in Taiwan.

In order to address some of these issues, this study adopts a multi-site, prospective clinical follow-up design. It aims at establishing a research network for examining MMT outcome, developing standardized MMT outcome assessment instruments and procedures, and identifying predictors of MMT outcome. The findings may contribute to the better understanding of the characteristics of opioid addicts, the effectiveness of MMT and remaining service needs for opioid addicts in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Be fulfilling the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of opiate dependence.
* Be agree to and capable of signing informed consent form that has been approved by an Institution Review Board.

Exclusion Criteria:

* Have ever participated in the study at one of the collaborative hospitals/clinics.
* Be expecting to discontinue methadone treatment for any reason (leaving the methadone clinic's geographic area, pending legal action, etc.) in the following 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heroin-addicted patients who seek help for methadone maintenance treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chang Wang, M.D.,M.Sc., Principal Investigator — National Health Research Institutes, Taiwan
Locations (7):
- Taiwan (7):
  - Departments of Psychiatry, Wei-Gong Memorial Hospital, Miaoli
  - Departments of Psychiatry, China Medical University and Hospital, Taichung
  - Departments of Psychiatry, Far-Eastern Memorial Hospital, Taipei
  - Departments of Psychiatry, Taipei City Hospital Song-De Campus, Taipei
  - Departments of Psychiatry, Taipei City Hospital Yang-Ming Campus, Taipei
  - Departments of Psychiatry, En-Chu-Kong Hospital, Taipei County
  - Departments of Psychiatry, Tao-yuan Psychiatric Center, Taoyuan District